CLINICAL TRIAL: NCT05027178
Title: Phenotypic Comparison of Ischemic and Hemorrhagic Stroke Patients Receiving Chiropractic Care Post-rehabilitation
Brief Title: Stroke Patients Receiving Chiropractic Care Post-rehabilitation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study is being reformatted and will have a different protocol for the relaunch.
Sponsor: Life University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: I-0014
Record Dates: First submitted 2021-08-27; First posted 2021-08-30 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data analysis - single blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chiropractic care for Ischemic Stroke Patients (Experimental): 12 weeks of full spine chiropractic care will be provided to patient. Patients may be asked to present one- two times per week.
  Interventions: Other: Chiropractic Care
- Chiropractic care for Hemorrhagic Stroke Patients (Experimental): 12 weeks of full spine chiropractic care will be provided to patient. Patients may be asked to present one- two times per week.
  Interventions: Other: Chiropractic Care

INTERVENTIONS:
Other: Chiropractic Care — Chiropractic care on stroke participants

SUMMARY:
The Life University Center for Chiropractic Research is conducting a research study to better understand how 12-weeks of chiropractic care differentially affects the post-rehabilitation brain electrical patterns and body movement patterns of individuals who have experienced hemorrhagic versus ischemic stroke The study will involve visits to the Life University Center for Chiropractic Research (CCR) in midtown Atlanta. During the 12 weeks of focused care, chiropractic visits could be several times a week depending on the care plan. In addition to the chiropractic care, individuals will receive a physical examination and three follow-up assessments. The assessments in the CCR will include a non-invasive evaluation of the brain wave patterns using electroencephalography (EEG), completion of a few surveys, a balance assessment and a movement assessment. Qualified individuals will receive study treatment and care at no cost.

ELIGIBILITY:
Inclusion Criteria:

* Post stroke rehabilitation

Exclusion Criteria:

* Not experienced sub-arachnoid bleeding within the last 4 weeks, fractures or trauma to the skull, pregnancy, or progressive RA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Stroke Impact Scale Survey | Baseline
  Disease specific self-report questionnaire that evaluates disability and health related quality of life post stroke.
Stroke Impact Scale Survey | 4 weeks
  Disease specific self-report questionnaire that evaluates disability and health related quality of life post stroke.
Stroke Impact Scale Survey | 8 weeks
  Disease specific self-report questionnaire that evaluates disability and health related quality of life post stroke.
Stroke Impact Scale Survey | 12 weeks
  Disease specific self-report questionnaire that evaluates disability and health related quality of life post stroke.
Resting State Electroencephalography | Baseline
  EEG assessment
Resting State Electroencephalography | 4 weeks
  EEG assessment
Resting State Electroencephalography | 8 weeks
  EEG assessment
Resting State Electroencephalography | 12 weeks
  EEG assessment
Kinematic Assessment of Performance on finger to nose test | Baseline
  Assessment to measure of dysmetria
Kinematic Assessment of Performance on finger to nose test | 4 weeks
  Assessment to measure of dysmetria
Kinematic Assessment of Performance on finger to nose test | 8 weeks
  Assessment to measure of dysmetria
Kinematic Assessment of Performance on finger to nose test | 12 weeks
  Assessment to measure of dysmetria

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sullivan, DC, PhD, Principal Investigator — Life Univeristy
Locations (1):
- Life University Center for Chiropractic Research, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No